CLINICAL TRIAL: NCT00202475
Title: Collection of Autologous Blood Products by Double Erythrocytapheresis - Cost Effectiveness Study
Brief Title: Collection of Autologous Blood Products by Double Erythrocytapheresis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Atrium Medical Center (Other); Maasland Hospital (Other)
Responsible Party: Dr. Wim de Kort PhD, Sanquin Blood BankDivision South-east
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPO-C-02-15
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Pre Operative Autologous Donation
Keywords: Dubble eerythrocytapheresis
MeSH Terms: interventions — Blood Component Removal; Blood Donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: eythrocytapheresis
- 2 (Active Comparator)
  Interventions: Procedure: whole blood collection

INTERVENTIONS:
Procedure: eythrocytapheresis — machinal collection of erythrocytes
  Other Names: apheresis
  Arms: 1
Procedure: whole blood collection — collection of whole blood
  Other Names: blood donation
  Arms: 2

SUMMARY:
The project will determine the advantages of double erythrocytapheresis in the collection of preoperative autologous erythrocytes as compared to the standard collections of whole blood. The study will assess the total reduction in the number of procedures required to obtain the preoperative units ordered by the surgeon. Also, successfulness of erythrocytaphereses versus classical whole blood collection for these patients will be compared.

DETAILED DESCRIPTION:
The project will determine the advantages of double erythrocytapheresis in the collection of preoperative autologous erythrocytes as compared to the standard collections of whole blood. The study will assess the total reduction in the number of procedures required to obtain the preoperative units ordered by the surgeon. Also, successfulness of erythrocytaphereses versus classical whole blood collection for these patients will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery

Exclusion Criteria:

* Malignancies
* Severe arrhythmias
* Congestive heart failure
* Recent angina
* Epileptic seizures in the last 3 months before collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-09; Primary Completion 2006-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
decline in Hemoglobine levels | surgery

SECONDARY OUTCOMES:
Storage parameters- ATP | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Eva Rombout, MD, Principal Investigator — Sanquin Research and Blood Bank Divisions
Locations (2):
- Netherlands (2):
  - Sanquin Bloodbank, Maastricht, Limburg
  - Sanquin Blood Bank Southeast Region, Maastricht